CLINICAL TRIAL: NCT02076893
Title: A Comparison of Postoperative Tramadol/Gabapentin/Ibuprofen Versus Tramadol/Placebo/Ibuprofen in Children Undergoing Tonsillectomy
Brief Title: Postoperative Tramadol/Gabapentin/Ibuprofen Versus Tramadol/Placebo/Ibuprofen
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis results indicated need to recruit beyond scope of budget.
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHC-IRGP-Gaba
Record Dates: First submitted 2014-02-11; First posted 2014-03-04 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Pain
Keywords: Tonsillectomy; Pain management; Pediatrics
MeSH Terms: conditions — Pain; Agnosia | interventions — Gabapentin; Tramadol; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tramadol/gabapentin/ibuprofen (Active Comparator): (A) Scheduled tramadol 1mg/kg Q6h [max. 50mg] for 5 days; plus tramadol 1mg/kg Q6h PRN [max. 50mg] for 5 days (B) Scheduled gabapentin 3 mg/kg [max 150 mg] Q6h for 5 days (C) PRN ibuprofen 10 mg/kg [max. 500 mg] Q6h PRN
  Interventions: Drug: gabapentin; Drug: Tramadol; Drug: Ibuprofen
- Tramadol/placebo/ibuprofen (Placebo Comparator): (A) Scheduled tramadol 1mg/kg Q6h [max. 50mg] for 5 days; plus tramadol 1mg/kg Q6h PRN [max. 50mg] for 5 days (B) Scheduled placebo of same volume Q6h for 5 days (C) PRN ibuprofen 10 mg/kg [max. 500 mg] Q6h PRN
  Interventions: Drug: Tramadol; Drug: Ibuprofen; Drug: Placebo

INTERVENTIONS:
Drug: gabapentin — The active comparator arm will receive gabapentin as per dosing specifics listed in the study arm description.
  Other Names: Neurontin
  Arms: Tramadol/gabapentin/ibuprofen
Drug: Tramadol — Both study arms will receive tramadol per dosing details listed in the study arm descriptions.
  Other Names: Ultram
Drug: Ibuprofen — Both study arms will receive as needed (PRN) ibuprofen to take home.
  Other Names: Advil; Motrin
Drug: Placebo — Simple syrup suspension
  Arms: Tramadol/placebo/ibuprofen

SUMMARY:
Tonsillectomy is the most common pediatric surgical procedure performed in the US, with over 530,000 procedures performed annually in children under 15 years (Baugh et al., 2011). The postoperative period can be particularly painful. A recent clinical consensus acknowledges there is no standard analgesic protocol, and calls for further research comparing postoperative pain medications (Baugh et al., 2011). Tramadol was found to be as effective as codeine with few reported side effects in a recent double-blinded, controlled trial conducted by the investigators at Children's Hospitals and Clinics (CHC), and it is currently being prescribed in the postoperative setting. However, despite its effectiveness for pain control, there were some children that continued to report pain during the 10-day follow-up period. In response, the investigators will conduct a randomized, double-blinded controlled trial to determine whether or not adding scheduled gabapentin to a scheduled tramadol + "as needed" (PRN) ibuprofen regimen provides better pain control than tramadol + ibuprofen PRN alone during the post-tonsillectomy period. Using a 10-day take-home diary, caregivers will be asked to record daily information about their child's postoperative pain and other core outcomes and domains as recommended in the recent consensus statement put forth by the Pediatric Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) (McGrath et al., 2008). This study will offer new information regarding the efficacy and side effects associated with adding scheduled gabapentin to a postoperative pain management protocol in a pediatric population.

DETAILED DESCRIPTION:
Hypotheses

H1: Children who receive scheduled tramadol 1mg/kgQ6h with scheduled gabapentin (3 mg/kg/q6h dose) and PRN ibuprofen will experience better pain relief than children who receive scheduled tramadol 1mg/kgQ6h with PRN ibuprofen following tonsillectomy.

H2: Children who receive scheduled tramadol 1mg/kgQ6h with scheduled gabapentin and PRN ibuprofen will report fewer side effects than children who receive scheduled tramadol 1mg/kgQ6h with PRN ibuprofen following tonsillectomy.

This prospective study will include children ages 4 to 15 that are scheduled to undergo a tonsillectomy (with or without adenoidectomy) procedure at CHC's Minneapolis campus with one of the three Children's Ear, Nose, Throat and Facial Plastic Surgery surgeons. The three surgeons will perform the same standardized surgical technique. The study will be prospective, randomized, and double-blinded. Neither the patient /caregiver(s) nor the person(s) evaluating the patient postoperatively will know whether the patient was assigned to Group 1 or Group 2. A random numbers list will be generated to assign sequential patients to Group 1 or Group 2 in order to eliminate selection bias due to group assignment or post-operative evaluation.

To minimize any potential risks associated with either tramadol or gabapentin when administered to obese children (i.e, children at the 85th percentile BMI or higher) the medication dose will be capped at a rate representing the 85th percentile for the child's age, sex and height.

Caregivers will be advised to administer the scheduled tramadol for five days along with scheduled gabapentin (or placebo) for five days. PRN doses of ibuprofen may be administered throughout the 10-day study period. For postoperative days 6-10, both groups will be advised to switch to a PRN regimen of ibuprofen and tramadol.

Caregivers will be advised NOT to administer any study medication if the child shows signs of over-sedation (respiratory rate lower than normal, slurred speech, etc.) or vomiting as a result of the study drug, AND will be asked to call the Ear Nose & Throat group in case of severe pain and or side effects (24/7 contact information will be provided). If the patient displays signs of severe over-sedation (breathing rate less than 12 breaths/minute, difficulty or inability to be aroused) parents will be advised to call 911. If in doubt, the caregiver will be asked to call the 24/7 ENT group phone number.

For all adverse events that arise during the study period, both non-urgent and urgent, the first point of contact for families will be with Children's Ear Nose & Throat and Facial Plastic Surgery. If families contact Children's pharmacy with any questions related to dosing or side effects, pharmacy staff will either contact Children's Ear, Nose & Throat and Facial Plastic Surgery themselves or refer the family to do so. For severe adverse events (respiratory depression, over sedation, seizure, etc.) and/or the child is seen by a physician due to potential drug side effects, the pharmacist will be authorized to break the blind. If in doubt, the pharmacist can call Children's Ear, Nose & Throat and Facial Plastic Surgery for guidance.

Staff Assessment and Caregiver Diary

The following patient and clinical information will be collected by research staff: patient's age, gender, race, diagnosis (apnea or chronic tonsillitis), concomitant medication use, postoperative pain, and tonsil size rated on a scale of 1 to 4 (see Appendix I).

The choice of outcome domains and measures in this study is based on a consensus paper developed by the Pediatric Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (PedIMMPACT) expert panel (McGrath et al., 2008). Acute pain domains are included in the caregiver diary for this study.

A daily diary will be completed by the caregiver and will be used to track the patient's pain symptoms, side effects, adverse events, and recovery during the first 24 hours and ten days post-surgery. This diary was developed and modified based on feedback received for the diary used in the recent clinical trial (Friedrichsdorf, unpublished). In addition, the research coordinator will contact the caregiver every second day to collect the same data and insure that the diary is completed. The patient /caregiver data will be compared to responses provided during the telephone call in order to validate diary entries. Intensity of pain and discomfort due to pain will be measured utilizing several methods including: a validated pain scale, documentation of use of analgesics and rescue medications, waking from sleep, time to ability to eat solid food, and time to return to normal activity. Other outcome measures include: fluid intake, general satisfaction with treatment, and economic impact of recovery (e.g., need for additional outpatient care for throat and/or ear pain, bleeding, nausea, or poor eating).

In this study, pain self-assessment by the children and adolescents will include the Faces Pain Scale-Revised (FPS-R) (with anchors 0=no pain and 10=highest pain imaginable) for children ages 4-10 (Hicks et al., 2001), and NRS-11 (with anchors 0=no pain and 10 = highest pain imaginable) for children ages 11-15 (note: children age 8-10 years will be asked to choose either the FPS-R or NRS-11, as both scales are validated for use with children in this middle age range). The designated caregiver participating in the study will receive training on pain scale administration. The study coordinator or research associate will call caregivers every two days during the follow-up period to remind them to complete the diary and return it in the postage-paid envelope provided by research staff.

Data Requirements and Data Maintenance

All paper forms will be stored in a locked file cabinet located in the Pain and Palliative Care department office. Data will be entered into Excel on a secure, password-protected Children's server and will be exported to SPSS for analysis. The study coordinator will maintain all paper and electronic data.

Risks/Benefits

Risks There is no additional medical risk associated with post-surgical pain management above and beyond the usual risks. Neither tramadol nor gabapentin pose any known additional safety risk. However, because little has been published in the pediatric literature about these two medications and their application in the postoperative setting, the researchers will form a small Data and Safety Monitoring Committee comprised of Children's staff members who are not part of the study. This committee will be responsible for reviewing serious adverse events as requested by the researchers (e.g., pharmacist, pain expert, etc.). As with any study, there is a risk of loss of confidentiality due to the possibility that people outside the study (e.g., staff, other families) may become aware of the child's participation in the study. The researchers will make every effort to ensure patients' privacy through use of private rooms for all research-related activities. Paper research forms will be stored in the Pain and Palliative Care office in a locked file cabinet, and all electronic data will be stored on a password-protected file on the Children's server.

Benefits There is a possibility that children who receive tramadol plus gabapentin with PRN ibuprofen during the recovery period will report better pain control, fewer side effects, or both than the children who receive tramadol plus PRN ibuprofen only. Future children and their families may benefit from the knowledge gained from the study in terms of improved pain management during the post-tonsillectomy recovery period.

Analysis

Analysis Plan

The following outcomes will be measured at two, four and 24 hours post-surgery, and then daily for the duration of the follow-up period:

* Pain: Faces Pain Scale-Revised (FPS-R) or Numerical Rating Scale (NRS-11)
* Postoperative pain: Parents' Postoperative Pain Measure (PPPM)
* Pre/Postoperative medication use, including any rescue medications
* Patient- and caregiver-reported side effects
* Sleep: difficulty falling asleep or difficulty waking
* Fluid intake
* Number of patients requiring outpatient care for complications of tonsillectomy including, but not limited to: throat and/or ear pain, bleeding, nausea
* Parent global satisfaction with treatment, recorded as 0-10 (0=Very Dissatisfied to 10=Very Satisfied) on a visual analog scale.

Descriptive statistics will be used to describe the participants and measurement results including frequency distribution for categorical data such as gender and any sleep problem (Yes/No), and mean (standard deviation) or median (range) for continuous data such as age, fluid intake, pain intensity score and parent global satisfaction with their child's recovery.

The number of days with pain intensity score greater than 4 will be compared between the tramadol/ibuprofen group and tramadol/gabapentin/ibuprofen group using a two-sample t-test or Mann-Whitney test. The PPPM scores and parental global satisfaction with their child's recovery between two groups will be compared using the two-sample t-test or Mann-Whitney test as well. Eta correlation coefficients will be calculated to examine the relationship between PPPM score and the pain intensity score. Chi-square test or Fisher's exact test will be used to compare the categorical data between two groups such as percent of patients having any postoperative office visit due to pain/bleeding/nausea and any side effects happened during the postoperative 10 days. A logistic regression model will be fit with 'patients having >2 days of pain score of > 4' as the dependent variable and other factors such as patient age, procedure, medication as independent variables in order to identify clinical factors predictive of postoperative pain following tonsillectomy in children.

Sample Size

Group sample sizes of 30 and 30 achieve 80% power to detect a difference of 2 in days with pain score > 4 between the Tramadol group and the Gabapentin group with estimated group standard deviations of 2.7 and with a significance level of 0.05 using a two-sided two-sample t-test. Assuming a 20% dropout, at least 36 patients will be needed in each group. The researchers plan to enroll at least 80 parents.

Environment

The study will take place on Children's Minneapolis campus. Data will be stored in the Pain, Palliative and Integrative Medicine office, currently located in the Medical Doctor's Building. This study will make use of CHC's outpatient pharmacy services in order to ensure proper dispensing and blinding.

ELIGIBILITY:
Inclusion Criteria:

* Child must be scheduled to undergo tonsillectomy (with or without adenoidectomy)
* Child must be between the ages of 4 and 15 at the time of enrollment.
* Child and caregiver must be English-speaking
* The same caregiver (e.g., mother) must agree to complete all study assessments with child to ensure consistency

Exclusion Criteria:

* Child cannot self-assess pain due to conditions such as developmental delays, chromosomal abnormalities, or other syndromes
* Child had significant adverse effects to tramadol, gabapentin and/or ibuprofen in the past
* Child has a known underlying seizure disorder (not febrile seizure)
* Child has known underlying renal or liver dysfunction (with creatinine, aspartate aminotransferase /alanine aminotransferase, more than twice above normal value for age, respectively)
* Child is taking an selective serotonin reuptake inhibitor (SSRI), norepinephrine reuptake inhibitor (SNRI), monoamine oxidase inhibitor (MAOI) or tricyclic

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2014-03; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of scheduled tramadol (days 1-5) + PRN ibuprofen (days 1-10)+ PRN tramadol (days 6-10) VS. scheduled tramadol (days 1-5) + scheduled gabapentin (days 1-5) + PRN ibuprofen (days 1-10) + PRN tramadol (days 6-10) | 10-day post-tonsillectomy recovery period
  To compare the efficacy of scheduled tramadol + PRN ibuprofen/tramadol vs. scheduled tramadol + scheduled gabapentin + PRN ibuprofen/tramadol for pain management during the post-tonsillectomy recovery period. Efficacy will be measured through daily collection of three pain scores (FACES or numeric; 0-10 rating): "pain right now," "typical pain over the past 24 hours," and "worst pain in the past 24 hours." Efficacy will also be measured daily with: 1) the Parents' Postoperative Pain Measure, 2) the number of times "as needed" medication is given by parents, 3) sleep quality, and 4) global satisfaction with pain management and recovery (on day 10 only). All efficacy measures will be recorded in a take-home diary by parents for 10 days postoperatively.

SECONDARY OUTCOMES:
Side effects of scheduled tramadol (days 1-5) + PRN ibuprofen (days 1-10)+ PRN tramadol (days 6-10) VS. scheduled tramadol (days 1-5) + scheduled gabapentin (days 1-5) + PRN ibuprofen (days 1-10) + PRN tramadol (days 6-10) | 10-day post-tonsillectomy recovery period
  To evaluate the side effects of scheduled tramadol + PRN ibuprofen/tramadol vs. scheduled tramadol + scheduled gabapentin + PRN ibuprofen/tramadol during the post-tonsillectomy recovery period. Safety will be measured through use of a daily take-home diary that the parents fill out, and through phone calls made to parents by the study coordinator every two days during the 10-day recovery period. Specifically, parents will document, on a daily basis, number and occurence of any side effects (e.g., vomiting, dizziness), number of doctor and emergency room visits, length of stay in days (if applicable), and the purpose and location of any medical visits.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Friedrichsdorf, MD, Principal Investigator — Childrens's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided